CLINICAL TRIAL: NCT04636671
Title: Randomized Controlled Trial of Methylprednisolone Versus Dexamethasone in COVID-19 Pneumonia (MEDEAS Trial)
Brief Title: Methylprednisolone vs. Dexamethasone in COVID-19 Pneumonia (MEDEAS RCT)
Acronym: MEDEAS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Trieste (Other)
Collaborators: Centro di Riferimento Oncologico - Aviano (Other); National Institute for the Infectious Diseases (L. Spallanzani) - Rome (Unknown)
Responsible Party: Principal Investigator, Confalonieri Marco, MD, Professor, University of Trieste
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEDEAS1
Record Dates: First submitted 2020-11-18; First posted 2020-11-19 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Covid19; Viral Pneumonia Human Coronavirus; Severe Acute Respiratory Syndrome
Keywords: Methylprednisolone; Dexamethasone; COVID-19; Pneumonia
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome; Pneumonia | interventions — Methylprednisolone; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Open-label, randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methylprednisolone (Experimental): A. On day 1, loading dose of methylprednisolone (MP) 80 mg IV in 30 minutes, promptly followed by continuous infusion of MP 80 mg/day in 240 mL of normal saline at 10 mL/h.
  B. From day 2 to day 8: infusion of MP 80 mg/day in 240 mL of normal saline at 10 mL/h.
  C. From day 9 and beyond:
  1. If not intubated patient and PaO2/FiO2 > 200, taper to MP 20 mg IV in 30 minutes three times a day for 3 days, then MP 20 mg IV twice daily for 3 days, then MP 20 mg IV once daily for 2 days, then switch to MP 16 mg/day PO for 2 days, then MP 8mg/day PO for 2 days, then MP 4mg/day PO for 2 days;
  2. If intubated patient or PaO2/FiO2 <= 200 with at least 5 cmH2O CPAP, continue infusion of MP 80 mg/day in 240 mL of normal saline at 10 mL/h until PaO2/FiO2 > 200 then taper as in a)
  Interventions: Drug: Methylprednisolone
- Dexamethasone (Active Comparator): A. Dexamethasone (DM) 6 mg IV in 30 minutes or PO from day 1 to day 10 or until hospital discharge (if sooner).
  B. After day 10 study treatment is interrupted.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Methylprednisolone — Per-protocol methylprednisolone administration and tapering (see arm description)
  Arms: Methylprednisolone
Drug: Dexamethasone — Per-protocol dexamethasone administration (see arm description)
  Arms: Dexamethasone

SUMMARY:
Low-dose glucocorticoid treatment is the only intervention shown to significantly reduce mortality in cases of COVID-19 pneumonia requiring oxygen supplementation or ventilatory support. In particular, a large UK randomized controlled trial (RECOVERY trial) demonstrated the efficacy of dexamethasone at a dosage of 6mg/day for 10 days in reducing mortality compared to usual therapy, with a greater impact on patients requiring mechanical ventilation (36% reduction) or oxygen therapy (18% reduction) than on those who did not need respiratory support (doi: 10.1056/NEJMoa2021436). However, there is still paucity of information guiding glucocorticoid administration in severe pneumonia/ARDS and no evidence of the superiority of a steroid drug -nor of a therapeutic scheme- compared to the others, which led to a great heterogeneity of treatment protocols and misinterpretation of available findings. In a recent longitudinal observational study conducted in Italian respiratory high-dependency units, a protocol with prolonged low-dose methylprednisolone demonstrated a 71% reduction in mortality and the achievement of other secondary endpoints such as an increase in ventilation-free days by study day 28 in a subgroup of patients with severe pneumonia and high levels of systemic inflammation (doi: 10.1093/ofid/ofaa421). The treatment was well tolerated and did not affect viral shedding from the airways. In light of these data, the present study aims to compare the efficacy of a methylprednisolone protocol and that of a dexamethasone protocol based on previous evidence in increasing survival by day 28, as well as in reducing the need and duration for mechanical ventilation, among hospitalized patients requiring noninvasive respiratory support (oxygen supplementation and/or noninvasive ventilation).

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and sign the informed consent
2. SARS-CoV-2 positive on at least one upper respiratory swab or bronchoalveolar lavage
3. PaO2 <= 60 mmHg or SpO2 <= 90% or on oxygen therapy (any), CPAP or NPPV at randomization
4. Age >= 18 years old at randomization

Exclusion Criteria:

1. On invasive mechanical ventilation (either intubated or tracheostomized)
2. Heart failure as the main cause of acute respiratory failure
3. On long-term oxygen or home mechanical ventilation
4. Decompensated liver cirrhosis
5. Immunosuppression (i.e., cancer on treatment, post-organ transplantation, HIV-positive, on immunosuppressant therapy)
6. On chronic steroid therapy or other immunomodulant therapy (e.g., azathioprine, methotrexate, mycophenolate, convalescent/hyperimmune plasma)
7. Chronic renal failure with dialysis dependence
8. Progressive neuro-muscular disorders
9. Cognitively impaired, dementia or decompensated psychiatric disorder
10. Quadriplegia/Hemiplegia or quadriparesis/hemiparesis
11. Do-not-resuscitate order
12. Participating in other clinical trial including experimental compound with proved or expected activity against SARS-CoV-2 infection
13. Any other condition that in the opinion of the investigator may significantly impact with patient's capability to comply with protocol intervention
14. Refuse to participate in the study or absence of signed informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 690 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-05-04 (Actual)

PRIMARY OUTCOMES:
Survival | 28 days
  Survival proportion at 28 days in both arms

SECONDARY OUTCOMES:
Reduction in the need for mechanical ventilation | 28 days
  Number of days free from mechanical ventilation (either noninvasive or invasive) by study day 28 in both arms
Length of hospitalization | From date of randomization until the date of hospital discharge, assessed up to 60 days
  Number of days of hospitalization for patients discharged alive in both arms
Need for tracheostomy | Day 28
  Proportion of patients requiring tracheostomy in both arms
Reduction in systemic inflammation markers | Day 3, 7 and 14
  C-reactive protein level (mg/L) at study day 3, 7 and 14 in both arms
Amelioration of oxygenation | Day 3, 7 and 14
  PaO2/FiO2 ratio (mmHg) at study day 3, 7 and 14 in both arms
Disease progression | Day 3, 7 and 14
  WHO clinical progression scale at study day 3, 7 and 14 in both arms

CONTACTS AND LOCATIONS:
Overall Officials: Marco Confalonieri, MD, Principal Investigator — University of Trieste
Locations (1):
- Marco Confalonieri, Trieste, TS, Italy

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results of this study after deidentification, as well as study protocol, statistical analysis plan, informed consent form, clinical study report and analytic code will be made available to Researchers who provide a written proposal for their purposes. Proposals must be submitted to the study PI or co-PI up to 36 months following article publication. Requestors must sign a data access agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 36 months following article publication

REFERENCES:
- [Background] RECOVERY Collaborative Group; Horby P, Lim WS, Emberson JR, Mafham M, Bell JL, Linsell L, Staplin N, Brightling C, Ustianowski A, Elmahi E, Prudon B, Green C, Felton T, Chadwick D, Rege K, Fegan C, Chappell LC, Faust SN, Jaki T, Jeffery K, Montgomery A, Rowan K, Juszczak E, Baillie JK, Haynes R, Landray MJ. Dexamethasone in Hospitalized Patients with Covid-19. N Engl J Med. 2021 Feb 25;384(8):693-704. doi: 10.1056/NEJMoa2021436. Epub 2020 Jul 17. PMID 32678530
- [Background] Arabi YM, Chrousos GP, Meduri GU. The ten reasons why corticosteroid therapy reduces mortality in severe COVID-19. Intensive Care Med. 2020 Nov;46(11):2067-2070. doi: 10.1007/s00134-020-06223-y. Epub 2020 Oct 7. No abstract available. PMID 33026460
- [Background] WHO Rapid Evidence Appraisal for COVID-19 Therapies (REACT) Working Group; Sterne JAC, Murthy S, Diaz JV, Slutsky AS, Villar J, Angus DC, Annane D, Azevedo LCP, Berwanger O, Cavalcanti AB, Dequin PF, Du B, Emberson J, Fisher D, Giraudeau B, Gordon AC, Granholm A, Green C, Haynes R, Heming N, Higgins JPT, Horby P, Juni P, Landray MJ, Le Gouge A, Leclerc M, Lim WS, Machado FR, McArthur C, Meziani F, Moller MH, Perner A, Petersen MW, Savovic J, Tomazini B, Veiga VC, Webb S, Marshall JC. Association Between Administration of Systemic Corticosteroids and Mortality Among Critically Ill Patients With COVID-19: A Meta-analysis. JAMA. 2020 Oct 6;324(13):1330-1341. doi: 10.1001/jama.2020.17023. PMID 32876694
- [Background] Meduri GU, Annane D, Confalonieri M, Chrousos GP, Rochwerg B, Busby A, Ruaro B, Meibohm B. Pharmacological principles guiding prolonged glucocorticoid treatment in ARDS. Intensive Care Med. 2020 Dec;46(12):2284-2296. doi: 10.1007/s00134-020-06289-8. Epub 2020 Nov 4. PMID 33150472
- [Background] Salton F, Confalonieri P, Meduri GU, Santus P, Harari S, Scala R, Lanini S, Vertui V, Oggionni T, Caminati A, Patruno V, Tamburrini M, Scartabellati A, Parati M, Villani M, Radovanovic D, Tomassetti S, Ravaglia C, Poletti V, Vianello A, Gaccione AT, Guidelli L, Raccanelli R, Lucernoni P, Lacedonia D, Foschino Barbaro MP, Centanni S, Mondoni M, Davi M, Fantin A, Cao X, Torelli L, Zucchetto A, Montico M, Casarin A, Romagnoli M, Gasparini S, Bonifazi M, D'Agaro P, Marcello A, Licastro D, Ruaro B, Volpe MC, Umberger R, Confalonieri M. Prolonged Low-Dose Methylprednisolone in Patients With Severe COVID-19 Pneumonia. Open Forum Infect Dis. 2020 Sep 12;7(10):ofaa421. doi: 10.1093/ofid/ofaa421. eCollection 2020 Oct. PMID 33072814
- [Background] WHO Working Group on the Clinical Characterisation and Management of COVID-19 infection. A minimal common outcome measure set for COVID-19 clinical research. Lancet Infect Dis. 2020 Aug;20(8):e192-e197. doi: 10.1016/S1473-3099(20)30483-7. Epub 2020 Jun 12. PMID 32539990
- [Background] Dimairo M, Pallmann P, Wason J, Todd S, Jaki T, Julious SA, Mander AP, Weir CJ, Koenig F, Walton MK, Nicholl JP, Coates E, Biggs K, Hamasaki T, Proschan MA, Scott JA, Ando Y, Hind D, Altman DG; ACE Consensus Group. The Adaptive designs CONSORT Extension (ACE) statement: a checklist with explanation and elaboration guideline for reporting randomised trials that use an adaptive design. BMJ. 2020 Jun 17;369:m115. doi: 10.1136/bmj.m115. PMID 32554564
- [Derived] Reccardini N, Confalonieri M, Ruaro B, Confalonieri P, Da Re B, Rocca A, Salton F. Early C-reactive protein reduction predicts survival in COVID-19 severe pneumonia treated with glucocorticoids. BMC Pulm Med. 2025 Sep 30;25(1):436. doi: 10.1186/s12890-025-03874-9. PMID 41029298
- [Derived] Salton F, Confalonieri P, Centanni S, Mondoni M, Petrosillo N, Bonfanti P, Lapadula G, Lacedonia D, Voza A, Carpene N, Montico M, Reccardini N, Meduri GU, Ruaro B; MEDEAS Collaborative Group; Confalonieri M; MEDEAS Collaborative Group; Citton GM, Lapadula G, Bozzi C, Tavano S, Pozzan R, Andrisano AG, Jaber M, Mari M, Trotta L, Mondini L, Barbieri M, Ruggero L, Antonaglia C, Soave S, Torregiani C, Bogatec T, Baccelli A, Nalesso G, Re B, Pavesi S, Barbaro MPF, Giuliani A, Ravaglia C, Poletti V, Scala R, Guidelli L, Golfi N, Vianello A, Achille A, Lucernoni P, Gaccione AT, Romagnoli M, Fraccaro A, Malacchini N, Malerba M, Ragnoli B, Zamparelli AS, Bocchino M, Blasi F, Spotti M, Miele C, Piedepalumbo F, Barone I, Baglioni S, Dodaj M, Franco C, Andrani F, Mangia A, Mancini A, Carrozzi L, Rafanelli A, Casto E, Rogliani P, Ora J, Carpagnano GE, Di Lecce V, Tamburrini M, Papi A, Contoli M, Luzzati R, Zatta M, Di Bella S, Caraffa E, Francisci D, Tosti A, Pallotto C, De Rosa FG, Pecori A, Franceschini M, Carlin M, Orsini V, Spolti A, Inannace M, Santantonio T, Meli R, Sauro S, Fedeli C, Mangini E, Biolo G, Nunnari A, Pietrangelo A, Corradini E, Bocchi D, Boarini C, Zucchetto A, Lanini S. Prolonged higher dose methylprednisolone versus conventional dexamethasone in COVID-19 pneumonia: a randomised controlled trial (MEDEAS). Eur Respir J. 2023 Apr 20;61(4):2201514. doi: 10.1183/13993003.01514-2022. Print 2023 Apr. PMID 36356972